CLINICAL TRIAL: NCT00897455
Title: Genetic Modifiers of BRCA1/BRCA2-Related Breast Cancer Risk in BRCA1/BRCA2 Mutation Carriers - CIMBA 5
Brief Title: Studying Breast Cancer Risk in Women Who Are BRCA1/BRCA2 Mutation Carriers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000598427; GOG-8008
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Breast Cancer
Keywords: breast cancer; BRCA1 mutation carrier; BRCA2 mutation carrier
MeSH Terms: conditions — Breast Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: mutation analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Studying samples of DNA in the laboratory from women who are BRCA1/BRCA2 mutation carriers may help doctors learn more about cancer and identify biomarkers related to cancer.

PURPOSE: This research study is looking at breast cancer risk in women who are BRCA1/BRCA2 mutation carriers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify potential genetic modifiers of breast cancer risk by contributing data and genetic information obtained from women who are BRCA1/BRCA2 mutation carriers enrolled in clinical trial GOG-0199 to an international consortium of clinical cancer genetics investigators (CIMBA).

OUTLINE: This is a multicenter study. Patients are stratified by study, country of residence, ethnicity, and birth cohort. Joint analyses of BRCA1 and BRCA2 mutation carriers are further stratified by mutation.

Previously collected DNA samples are analyzed for genetic variants in selected candidate genes (rs16942 in BRCA1, rs2237060 in RAD50, "SNP3", and rs2241193 in IGFBP5). The single nucleotide polymorphism (SNP) data from this study and selected demographic, clinical, and epidemiological data obtained from the baseline questionnaire administered in the GOG-0199 study are submitted to the Consortium of Investigators of Modifiers of BRCA-Associated Cancer (CIMBA) Central Database. The epidemiological and SNP data contributed to the Central Database are then distributed to the investigators responsible for analysis of a particular SNP or set of SNPs from a candidate gene or genetic pathway.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Known positive BRCA1/BRCA2 mutation carrier
* With or without a personal history of breast cancer prior to enrollment in clinical trial GOG-0199
* Currently enrolled in clinical trial GOG-0199 AND meets the following criteria:

  * Completed baseline questionnaire (BQ-199)
  * Provided information on prior breast cancer history, including date of diagnosis
  * Provided complete data from the DNA analysis on the genetic variants of interest
  * Signed an approved informed consent and authorization permitting release of personal health information
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Identification of potential genetic modifiers of breast cancer risk

CONTACTS AND LOCATIONS:
Overall Officials: Mark H. Greene, MD, Study Chair — Clinical Genetics Branch; Michael Birrer, MD, PhD — NCI - Cell and Cancer Biology Branch; Phuong Mai, MD — Clinical Genetics Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States